CLINICAL TRIAL: NCT02900716
Title: A Phase Ia/Ib Study of a Novel BTK Inhibitor, DTRMWXHS-12, and Combination Products, DTRM-505 and DTRM-555, in Patients With Chronic Lymphocytic Leukemia or Other B-cell Lymphomas
Brief Title: Safety Study of BTK Inhibitor, DTRMWXHS-12, Used Singly or in Combination, in CLL and B-cell Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang DTRM Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D15-11094
Record Dates: First submitted 2016-08-18; First posted 2016-09-14 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-04

CONDITIONS: Chronic Lymphocytic Leukemia; B-Cell Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell | interventions — DTRMWXHS-12

ARMS (3):
- Phase Ia (Experimental): DTRMWXHS-12: oral capsules, daily x 21 days every 28 days
  Interventions: Drug: DTRMWXHS-12
- Phase Ib, DTRM-505 (Experimental): DTRMWXHS-12 oral capsules and everolimus oral tablets: daily x 21 days every 28 days
  Interventions: Drug: DTRM-505
- Phase Ib, DTRM-555 (Experimental): DTRMWXHS-12 and pomalidomide oral capsules, everolimus oral tablets:
  daily x 21 days every 28 days
  Interventions: Drug: DTRM-555

INTERVENTIONS:
Drug: DTRMWXHS-12 — DTRMWXHS-12
  Arms: Phase Ia
Drug: DTRM-505 — DTRMWXHS-12 and everolimus
  Arms: Phase Ib, DTRM-505
Drug: DTRM-555 — DTRMWXHS-12 and everolimus and pomalidomide
  Arms: Phase Ib, DTRM-555

SUMMARY:
This study will evaluate the safety, antitumor activity and preliminary pharmacokinetics of an investigational drug product, DTRMWXHS-12, in patients with chronic lymphocytic leukemia or other B-cell lymphomas. DTRMWXHS-12 will be evaluated as a single agent, and in combination.

This study will be conducted in two parts: phase Ia and Ib. Both parts will explore escalating doses of DTRMWXHS-12. The phase Ia study will evaluate DTRMWXHS-12 monotherapy. The phase Ib study will evaluate DTRMWXHS-12 combinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of chronic lymphocytic leukemia (CLL) or other B-cell neoplasms including small lymphocytic lymphoma (SLL), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL) and follicular B-cell non-Hodgkin's lymphoma (FL) who have no available approved therapies.
* Age > 18 years.
* Life expectancy greater than 12 weeks.
* Patients must have an ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1.
* Patients must provide written informed consent.
* Ability to swallow and retain capsules.
* Absence of uncontrolled intercurrent illnesses, including uncontrolled infections, cardiac conditions, or other organ dysfunctions.
* Women of child-bearing potential must have a negative serum or urine pregnancy test.
* Women of child-bearing potential must agree to use 2 reliable methods of contraception beginning 4 weeks prior to the initiation of treatment, during therapy, and for at least 4 weeks after the last drug administration.
* Men must agree to use a latex or synthetic condom during sexual contact with a pregnant female or a female who can become pregnant, for the duration of the study and for at least 4 weeks after the last drug administration, even if they have undergone a successful vasectomy.

Exclusion Criteria:

* Received previous chemotherapy, immunotherapy, radiotherapy or any other investigational therapy within 21 days or 5 half-lives for targeted therapies prior to this study entry.
* Patients with active infections requiring intravenous (IV) antibiotic/antiviral therapy are not eligible for entry onto the study until resolution of the infection; patients on prophylactic antibiotics, antifungals or antivirals are acceptable
* Pregnant or lactating individuals.
* Impaired hepatic or renal function as demonstrated by any of the following laboratory values:

  1. AST or ALT > 2.5 x ULN
  2. Total bilirubin > 1.5 x ULN (Patients with a history of Gilbert's syndrome may participate if total bilirubin is less than or equal to 1.5 x ULN and the AST/ALT and alkaline phosphatase meet the protocol-specified levels for eligibility)
  3. Alkaline phosphatase > 2.5 x ULN
  4. Glomerular filtration rate (GFR) < 50 mL/min, as assessed using the standard methodology at the investigating center (i.e. Cockroft-Gault), or serum creatinine > 1.5 x ULN
* INR > 1.5 or other evidence of impaired hepatic synthesis function.
* Persisting (> 8 weeks) severe pancytopenia due to hematologic disorder or due to previous therapy rather than disease (ANC < 0.5 x 109/L or platelets < 30 x 109/L) - to be confirmed via bone marrow biopsy, as part of normal clinical care, prior to signing of consent.
* Previous allogeneic bone marrow transplant are restricted, unless there is no evidence of acute or chronic graft versus host disease.
* CNS involvement with malignancy.
* Current malignancies of another type, with the exception of adequately treated in situ cervical cancer and basal cell skin cancer, squamous cell carcinoma of the skin or other malignancies with no evidence of disease for 2 years or more.
* Known history of HIV, HBV or HCV infection.
* Documented or known bleeding disorder.
* Requirement for anticoagulation treatment that increases INR or aPTT above the normal range (low molecular weight heparin and heparin line flush allowed).
* Patient is receiving any azole.
* Patients with a significant cardiovascular disease or condition, including:

  * Myocardial infarction within 6 months of study entry
  * NYHA Class III or IV heart failure, or reduced LVEF <50%
  * Uncontrolled dysrhythmias or poorly controlled angina.
  * History of serious ventricular arrhythmia (VT or VF, ≥ 3 beats in a row) and/or risk factors (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
  * Baseline prolongation of QT/QTc interval (repeated demonstration of QTc ≥ 450 msec for men and 470 msec for women, or LVEF ≤ 40% by MUGA or ECHO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-09; Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Starting from date of first dose up to 30 days after last dose
  Safety and tolerability

SECONDARY OUTCOMES:
Plasma concentration over time | Days 1-28 (first treatment cycle)
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Wei He, Ph.D., Study Director — Zhejiang DTRM Biopharma
Locations (6):
- United States (6):
  - Mayo Clinic, Phoenix, Arizona
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania